CLINICAL TRIAL: NCT01310803
Title: A PHASE 3B, RANDOMIZED, OPEN-LABEL, MULTI-CENTER STUDY TO EVALUATE THE EFFICACY AND SAFETY OF MAINTENANCE THERAPY WITH VALRUBICIN VERSUS NO MAINTENANCE, IN SUBJECTS TREATED WITH VALRUBICIN INDUCTION FOR CARCINOMA IN SITU (CIS) OF THE BLADDER
Brief Title: Multi-center Study to Evaluate the Efficacy and Safety of Maintenance Therapy With Valrubicin Versus no Maintenance, in Subjects Treated With Valrubicin Induction for Carcinoma in Situ (CIS) of the Bladder
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: Endo Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EN3329-301
Record Dates: First submitted 2011-03-04; First posted 2011-03-09 (Estimated); Results first posted 2014-10-22 (Estimated); Last update posted 2017-10-05 (Actual); Status verified 2017-09

CONDITIONS: Carcinoma in Situ; Transitional Cell Carcinoma; Non-muscle Invasive Bladder Cancer
Keywords: Urinary Bladder Neoplasms; Neoplasms; Urologic Neoplasms; Urogenital Neoplasms; Neoplasms by Site; Urinary Bladder Diseases; Urologic Diseases; TURBT; Valstar
MeSH Terms: conditions — Carcinoma in Situ; Carcinoma, Transitional Cell; Non-Muscle Invasive Bladder Neoplasms; Urinary Bladder Neoplasms; Neoplasms; Urologic Neoplasms; Urogenital Neoplasms; Neoplasms by Site; Urinary Bladder Diseases; Urologic Diseases | interventions — valrubicin; Standard of Care

ARMS (2):
- Maintenance therapy (Experimental): Chemotherapeutic: EN3329-301 (VALSTAR)
  Interventions: Drug: VALSTAR - Maintenance Therapy
- No Maintenance (Standard of care) (Other): Subjects randomized to No Maintenance (Standard of Care) will not receive any additional intravesical therapy
  Interventions: Other: No Maintenance treatment ( Standard of Care)

INTERVENTIONS:
Drug: VALSTAR - Maintenance Therapy — Treatment phase - 10 monthly intravesical installations starting 10 to 12 weeks after the beginning of induction. Follow-up phase
  Other Names: VALSTAR
  Arms: Maintenance therapy
Other: No Maintenance treatment ( Standard of Care) — Subjects randomized to No Maintenance (Standard of Care) will not receive any additional intravesical therapy
  Arms: No Maintenance (Standard of care)

SUMMARY:
This is a Phase 3b open-label, randomized, parallel-arm, multicenter study to evaluate the efficacy and safety of 10 monthly intravesical administrations of maintenance therapy with valrubicin following induction with valrubicin as compared to induction with valrubicin only in subjects with CIS of the bladder. The randomization will be 1:1 and subjects will be stratified by tumor type (CIS plus papillary disease vs. CIS only) and time from last bacillus Calmette-Guerin (BCG) failure (>1 year vs. <1 year).

ELIGIBILITY:
Inclusion Criteria:

1. Is 18 years of age and older at time of consent signing
2. Have histologically confirmed diagnosis of CIS of the bladder and received valrubicin induction therapy per the labeled indication.
3. Is disease-free following induction with intravesical valrubicin

   * Disease-free is defined as negative biopsy 10 to 12 weeks after the initiation of valrubicin induction
   * Valrubicin induction is defined as having received at least 3 of 6 weekly instillations
4. Is available for the duration of the study including follow-up (minimum 12 months from randomization)
5. Have an Eastern Cooperative Oncology Group (ECOG) performance status grade of 2 or less
6. Have no evidence of urothelial carcinoma involving the upper urinary tract or prostatic urethra (confirmed by extravesical work up, which may include radiological imaging and/or biopsy) within 6 months prior to randomization
7. Subjects (male and female) of child-bearing potential (including female subjects who are post-menopausal for less than 1 year) must be willing to practice abstinence or effective contraception (as defined by the investigator) during the study and be willing and able to continue contraception for 30 days after their last dose of study treatment
8. Is able to understand and give written informed consent

Exclusion Criteria:

1. Have current or previous history of muscle-invasive bladder cancer (MIBC)
2. Current or previous history of lymph node positive and/or metastatic bladder cancer
3. Have current evidence of pure squamous cell carcinoma, pure adenocarcinoma or pure undifferentiated carcinoma of the bladder
4. Is currently receiving systemic anti-cancer therapy (cytotoxic/cytostatic, immunotherapy or radiation)
5. Received treatment with an investigational agent within 30 days or 5 half-lives prior to randomization, whichever is longer
6. Received treatment with an intravesical chemotherapeutic agent (other than valrubicin or a single administration of mitomycin C post-transurethral resection of bladder tumor [TURBT]) within 3 months prior to randomization
7. Received treatment with valrubicin other than induction within 3 months prior to randomization
8. Have contraindication to valrubicin

   * Known hypersensitivity to anthracyclines or polyoxyl castor oil
   * Small bladder capacity, i.e. unable to tolerate a 75 mL instillation
   * Concurrent urinary tract infection
9. Absolute neutrophil count (ANC) <1000/µL and hemoglobin <10 g/dL
10. Have active cardiovascular disease such as myocardial infarction within the past 3 months, unstable angina pectoris, congestive heart failure (NYHA Class III or IV) or uncontrolled cardiac arrhythmia
11. Female subjects who are pregnant or lactating
12. Subjects of childbearing potential who are unwilling to practice abstinence or effective contraception (as defined by investigator) during the study and for 30 days after last dose of study treatment
13. Have current or history of documented or suspected malignancy of any organ system (diagnosed, treated or untreated) within the past 5 years (with the exception of adequately treated basal cell or squamous cell carcinoma of the skin and asymptomatic non-metastatic prostate cancer either previously successfully treated or currently under active surveillance or receiving hormone therapy only)
14. Is unable to tolerate intravesical administration or intravesical surgical manipulation (cystoscopy or biopsy) even with premedication
15. Have ongoing clinically significant active infections
16. Have any medical or psychiatric condition which, in the opinion of the investigator, would preclude the participant from adhering to the protocol or completing the trial per protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2011-05; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Philippe E Spiess, MD, MS, FACS, FRCS(C), Principal Investigator — H. Lee Moffitt Cancer Center and Research Institute
Locations (6):
- United States (6):
  - BCG Oncology, Phoenix, Arizona
  - The Urology Center of Colorado, Denver, Colorado
  - Urology Associates, Cumberland, Maryland
  - Delaware Valley Urology, Sewell, New Jersey
  - Associated Medical Professionals of New York, Syracuse, New York
  - Urologic Consultants of SE PA, Bala-Cynwyd, Pennsylvania

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Maintenance Therapy | No Maintenance (Standard of Care)
Started | 1 | 0
Completed | 0 | 0
Not Completed | 1 | 0
Not completed — Subject terminated by Sponsor | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Maintenance Therapy | No Maintenance (Standard of Care) | Total
Number analyzed (Participants) | 1 | 0 | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 |  | 0
  Between 18 and 65 years | 0 |  | 0
  >=65 years | 1 |  | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 |  | 0
  Male | 1 |  | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 |  | 0
  Not Hispanic or Latino | 1 |  | 1
  Unknown or Not Reported | 0 |  | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 |  | 0
  Asian | 0 |  | 0
  Native Hawaiian or Other Pacific Islander | 0 |  | 0
  Black or African American | 0 |  | 0
  White | 1 |  | 1
  More than one race | 0 |  | 0
  Unknown or Not Reported | 0 |  | 0

OUTCOME MEASURES:

1. Primary Outcome: To Evaluate the Efficacy of Maintenance Therapy With Valrubicin After Induction With Valrubicin, as Compared to Induction With Valrubicin Only in Subjects With CIS of the Bladder.
Description: time interval from randomization to an event. An event is defined as tumor recurrence (any stage or grade), tumor progression to muscle-invasive bladder cancer (MIBC), metastatic bladder cancer or death from any cause, whichever occurs first. Tumor recurrence or progression must be documented by biopsy/transurethral resection of bladder tumor (TURBT).
Time Frame: 2 years
Population: No analysis completed due to limited enrollment (1 subject) prior to study termination.
Arm/Group | Maintenance Therapy | No Maintenance (Standard of Care)
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: To Evaluate the Safety and Tolerability of Maintenance Therapy With Valrubicin After Induction With Valrubicin, as Compared to Induction With Valrubicin Only in Subjects With CIS of the Bladder
Description: The occurrence of serious adverse events (SAEs), occurrence of local adverse reactions (LARs), results of vital signs, physical exams and laboratory test, and study discontinuation due to inability to complete valrubicin instillations
Time Frame: 2 years
Population: No analysis completed due to limited enrollment (1 subject) prior to study termination.
Arm/Group | Maintenance Therapy | No Maintenance (Standard of Care)
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Arm/Group | Maintenance Therapy | No Maintenance (Standard of Care)
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/0
Other Adverse Events (participants affected / at risk) | 0/1 | 0/0

LIMITATIONS AND CAVEATS:
This study was terminated early. Only one subject was enrolled. No study results were generated.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Institution and/or Principal Investigator shall not publish or present information related to the Study without prior written permission of Sponsor. Sponsor may withhold permission if a publication or presentation is in violation of other agreements, is not consistent with academic standards, is false or misleading, or is for commercial purposes.